CLINICAL TRIAL: NCT01723241
Title: A Randomized, Placebo-controlled, Double-blind, Multiple-ascending-dose Study to Assess the Safety and Tolerability of XAF5 Gel Applied to the Skin of Healthy Volunteers
Brief Title: Phase 1 Study of XAF5 Gel Applied to Skin of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XAF5 A1
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XAF5 (Experimental)
  Interventions: Drug: XAF5, concentration A; Drug: XAF5, concentration B; Drug: XAF5, concentration C
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XAF5, concentration A
  Arms: XAF5
Drug: XAF5, concentration B
  Arms: XAF5
Drug: XAF5, concentration C
  Arms: XAF5
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a study to assess the safety, tolerability, and pharmacokinetics of XAF5 Gel when applied to the skin of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Must understand and provide informed consent
* Skin upon which a reaction would be visible
* Body weight >= 70 kg

Exclusion Criteria:

* Any active skin disease
* History of skin hypersensitivity
* Clinically significant abnormality on physical exam, ECG, or laboratory tests
* Positive test for HIV, Hepatitis B, or Hepatitis C

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Singer, MD, PhD, Study Director — Topokine Therapeutics